CLINICAL TRIAL: NCT03992664
Title: A Pilot Randomized Controlled Study on the Effects of an Educational Training Program on Skin Reactions Induced by Chemotherapies, Epidermal Growth Factor Inhibitors (EGFRI) Treatments, and Immunotherapies.
Brief Title: Education Intervention in Patients with Rash Due to Epidermal Growth Factor Receptor (EGFR) Treatment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus University of Technology (Other)
Responsible Party: Principal Investigator, ELENI PAPOUI, NURSE, PhD (C), Cyprus University of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 0000-0001-5580-7256
Record Dates: First submitted 2019-06-15; First posted 2019-06-20 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2022-08

CONDITIONS: Consent Form; Lung Cancer; Colon Cancer; Pancreas Cancer; Head and Neck Cancer; Breast Cancer
Keywords: rash, photosensitivity, pruritus, educational, chemotherapy, EGFRI, immunotherapy
MeSH Terms: conditions — Lung Neoplasms; Colonic Neoplasms; Pancreatic Neoplasms; Head and Neck Neoplasms; Breast Neoplasms; Exanthema; Photosensitivity Disorders; Pruritus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): The patients in the experimental group follow the educational program once weekly, for 4 weeks.
  Interventions: Other: Educational training program
- NON-INTERVENTION (No Intervention): The usual information was provided to them

INTERVENTIONS:
Other: Educational training program — The training program will focus on four parameters: cleanliness, hydration, protection from external stimuli, and finally early detection of skin side effects.
  The re-evaluation of the skin as well as the repetition of the questionnaires will be done every week for 4 weeks.
  Arms: Experimental

SUMMARY:
The main adverse reaction of EGFR seen in patients is rash. EGFR treated patients have a 24-95% incidence of rash depending on the type of treatment they receive. Skin toxicity may occur in more than 80% of patients treated with cetuximab.

If a severe rash (Grade 3 or 4) occurs, a dose reduction or discontinuation of treatment may be required. Also, infections are the main secondary side effect caused by the rash.

The aim of the study is through a randomized clinical trial feasibility study to investigate the effectiveness of an educational intervention in patients receiving EGFRI therapy.

It will be randomly selected which patients will belong to the intervention group and who in the control group. The type of program involves educational intervention.

DETAILED DESCRIPTION:
In recent years, EGFRI (Epidermal Growth Factor Receptor Inhibitor) have evolved as effective anti-cancer drugs. They are distinguished in monoclonal antibodies (cetuximab and panitumumab) and EGFR (TKIs) kinase inhibitors gefitinib, erlotinib and lapatinib, where they are used in the treatment of colon, rectal, head and neck, lung, pancreas and of breast.

According to studies, the usual treatment for the prevention and treatment of skin rash refers to the use of antibiotics such as doxycycline, tetracycline and cortisone products such as hydrocortisone. It is also recommended to use moisturizing cream.

The study of Carmine P. et al., 2011 mentions the need to investigate educational measures for the rash due to EGFR treatment.

ELIGIBILITY:
1. Adult cancer patients (>18).
2. Patients who suffered with pruritus, or rash or photosensitivity, in the onset of the symptoms.
3. Willing to participate.
4. Ability to complete the questionnaires.
5. A performance status of two or less on the Eastern Cooperative Oncology Group (ECOG).
6. Patients with no pre-existing dermatological condition that may limit the interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Skin grades | 4 weeks
  Repeated measurements were taken weekly regarding the grade of rash, pruritus and photosensitivity.

SECONDARY OUTCOMES:
Functional health and wellbeing status | 4 weeks
  The SF-36 questionnaire (since week 0) and DLQI questionnaire (since week 1) were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: ANDREAS CHARALAMBOUS, PhD, Study Director — Cyprus University of Technology
Locations (1):
- Eleni Papoui, Larnaca, ATHIENOU, Cyprus

IPD SHARING:
Plan to Share IPD: No